CLINICAL TRIAL: NCT05785871
Title: Hypertension, Brain Clearance, and Markers of Neurodegeneration
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-05020073; 5R01NS104364-03 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Hypertension
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — In addition to the tests and goals described, participants' data, images, blood samples, cerebrospinal fluid and extracted DNA (Deoxyribonucleic acid) may, with the subject's permission, also be stored and used for current and future research purposes not outlined here. Blood samples are stored including whole blood, serum, plasma, red blood cells (erythrocytes) and white blood cells (leukocytes). Data stored will encompass all clinical, cognitive and imaging data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Untreated Hypertension: in office SBP ≥140 at two separate occasions and currently treated with antihypertensive medications (uncontrolled), or in office SBP ≥ 140 at two different occasions and no current treatment (untreated).
- Normotensive: in office SBP<140 mmHg, no treatment with antihypertensive medications
- Controlled Hypertension: in office SBP <140 and current treatment with antihypertensive medications

SUMMARY:
The purpose of this research study is to measure cerebrospinal fluid (CSF) clearance in subjects with and without high blood pressure. CSF cushions the brain from impact and carries waste products from the brain to the bloodstream. This process is known as clearance. Impaired removal of proteins from the aging brain causes their buildup and may contribute to an increased risk for Alzheimer's disease. It is also suspected that clearance may be related to the health of vessels carrying the blood throughout the brain. It is known that high blood pressure damages blood vessels and thus may impair clearance. In this project we will examine if having high blood pressure is related to impaired brain clearance and whether treating high blood pressure improves clearance and reduces buildup of Alzheimer's disease-related proteins.

Participants will be asked to undergo a medical examination, testing of memory, brain imaging (both magnetic resonance and positron emission tomography, and spinal tap at the beginning of the study and 1 -2 years later.

DETAILED DESCRIPTION:
Over 5 years the investigator will conduct a 24-month longitudinal study of 80 cognitively healthy subjects 60-80 years old, classified at baseline into the following groups: 1) Normotensive NT (n=20), 2) Controlled hypertension C-HTN (n=20), 3) Uncontrolled hypertension or Untreated hypertension UU-HTN (n=30).

For subjects in the NT and C-HTN groups this will be an observational longitudinal study with clinical, imaging and CSF (cerebrospinal fluid) assessment at baseline and 24 month follow-up, with 3 visits to monitor BP (blood pressure) in-between (both at the office and using home BP monitoring). Subjects in the UU-HTN group after having completed their baseline evaluation will be referred for a further evaluation of HTN (hypertension) and an intervention. Intervention: the initiation of treatment or treatment modification to achieve the SBP (systolic blood pressure) goal of <140 mmHg. Subjects will be referred to their physician or, in case they do not have one, to the study cardiologist for treatment according to current guidelines. Imaging at 0 and 24 month consist of MRI (magnetic resonance imaging) with ASL (arterial spin labeling) and brain clearance imaging using 18F-MK6240 PET (positron emission tomography). CSF assessment includes Aβ42 (amyloid beta 42), t-tau (total tau) and p-tau181 (tau phosphorylated at threonine 181).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 60-80 years old
* All subjects will speak English as their first language or demonstrate proficiency in English.
* All subjects will have normal cognition at baseline: a Clinical dementia rating CDR=0, Global deterioration Scale GDS <2
* For the HTN subjects: systolic HTN defined according to Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood pressure (JNC) 7 report. Specifically: Blood pressure in the ranges greater or equal to 140 mmHG, which is a mean of three seated BP readings on each of two or more office visits

Exclusion Criteria:

* Non-essential hypertension
* Diabetes
* Isolated diastolic hypertension
* Neurodegenerative disorders (i.e Parkinson disease)
* Dementia or Mild cognitive impairment at baseline
* Long life major depression. Baseline scores greater or equal to 20 on Beck Depression Inventory at baseline
* Long-life DSM-IV axis 1 disorders
* Mental retardation
* Substance abuse

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cognitively healthy, with and without hypertension, age 60-80, both men and women
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow | Baseline and up to 24 month follow up
  cerebral blood flow with arterial spin labeling MRI
Change in Brain Clearance | Baseline and up to 24 month follow up
  the rate of radiotracer removal from the brain ventricle after injection of MK-6240 images, measured with positron emission tomography
Change in total tau | Baseline and up to 24 month follow up
  total tau protein measured in cerebrospinal fluid
Change in amyloid 42 | Baseline and up to 24 month follow up
  amyloid 42 protein measured in cerebrospinal fluid
Change in cognitive performance | Baseline and up to 24 month follow up
  A composite score of tests assessing:
  Immediate and delayed memory (score ranges in parentheses):
  Craft Story immediate (0-44) and delayed recall (0-44), Guild battery immediate (0-21) and delayed recall (0-21) of paragraph and word pairs immediate (0-10) and delayed (0-10).
  Working memory:
  Number Span test forward (0-14) and backward (0-14)
  Naming:
  Verbal Naming Test (0-26).
  Attention:
  Trail Making Test part A (0-25)
  Executive functions:
  Trail Making Test Part B (score range 0-13) and Wisconsin Sorting Card Test (0-128).
  Verbal Fluency:
  Category Fluency: animals (0-30) and vegetables (0-30), category letters F (0-30) and L (0-30).
  Each test is transformed into normative z-score. For each domain the scores are expressed as a composite z-score of all the tests assessing a given domain. The score range from -3.0 - to +3.0 higher indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Glodzik, Principal Investigator — Weill Cornell MC
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participants data will be available after publication of final results.
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: Researchers who provide IRB-approved, methodologically sound proposal.